CLINICAL TRIAL: NCT05123287
Title: A Perspective, Self-control Study on the Progression of Carotid Plaques in Anti-PD-1 mAb Treated Tumor Patients by Artery Ultrasound Follow-up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-221
Record Dates: First submitted 2021-09-09; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Plaque, Atherosclerotic; Immune Checkpoint Inhibitors; Programmed Cell Death Protein 1 Inhibitor; Carotid Artery Plaque; Intimal Medial Thickness of Internal Carotid Artery
MeSH Terms: conditions — Plaque, Atherosclerotic; Carotid Stenosis; Carotid Intimal Medial Thickness 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: PD-1 immune checkpoint blockades — intravenous injection; frequency: 2-3 weeks/cycle; duration: 3 months

SUMMARY:
A Perspective, Self-control Study on the Progression of Carotid Plaques in Anti-PD-1 mAb Treated Tumor Patients by Artery Ultrasound Follow-up

DETAILED DESCRIPTION:
This is a perspective, self-controlled cohort study. This study aims to evaluate the effectiveness of anti-PD-1 mAbs (PD-1 immune checkpoint blockades) on atherosclerotic carotid plaques in those anti-PD-1 mAbs treated patients. The method for quantification and evaluation of atherosclerotic plaques are based on the: ① The mean intima-media thickness of the common carotid artery (Mean CCA thickness); ② The maximum intima-media thickness of the internal carotid artery (maximum ICA thickness); ③ Carotid plaque burden: by calculation of the plaque area of atherosclerotic plaques on the long axis direction of artery on the ultrasound images. By comparing the above-mentioned parameters at the same location of carotid artery in each patient when initiate the first-dose of anti-PD-1 mAbs therapy and 3 months post anti-PD-1 mAbs therapy. It is designed to assess the effectiveness of anti-PD-1 mAbs on the progression of carotid plaques.

ELIGIBILITY:
Inclusion Criteria:

1. The age of subjects are between 18-90 years old (including 18 and 90 years old);
2. All kinds of tumor diseases of subjects are acceptable;
3. All kinds of PD-1 immune checkpoint blockades or dosages are acceptable;
4. The subjects knew about the experiment and signed the informed consent voluntarily;
5. The subjects plan to receive PD-1 immune checkpoint blockades and potentially to be treated for over 3 months;
6. The subjects complicated with atherosclerotic carotid plaques.

Exclusion Criteria:

1. Subjects stop receiving or changing the PD-1 immune checkpoint blockades during follow-up;
2. Subjects are reluctant to continue to be involved in this study;
3. Known pregnant and lactating women;
4. The parameters (e.g., CCA intima-media, ICA intima-media or carotid plaque burden) could not be calculated because of the quality of ultrasound image;
5. Other situations that the researchers judged were not suitable for inclusion.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population are the PD-1 immune checkpoint blockade treated tumor patients from 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The mean intima-media thickness of the common carotid artery | 3 months
  It was measured over a segment of the common carotid artery that was 1 cm long, located approximately 0.5 cm below the carotid-artery bulb, and considered not to contain any plaque (i.e., not to have any perceivable protrusion of the artery wall into the lumen).
The maximum intima-media thickness of the internal carotid artery | 3 months
  It was defined as the greatest intima-media thickness in either the right or left internal carotid artery extending from the bulb to 1 cm above the carotid sinus, ascertained from a total of four views on each side.
Carotid plaque burden | 3 months
  Carotid plaque area measured by ultrasound (cross-sectional area of longitudinal views of all plaques seen) to quantify the increase or decrease of atherosclerotic carotid plaques.

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, MD, PhD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine at Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spence JD. Measurement of carotid plaque burden. JAMA Neurol. 2015 Apr;72(4):383-4. doi: 10.1001/jamaneurol.2014.3002. No abstract available. PMID 25686472
- [Background] O'Leary DH, Polak JF, Kronmal RA, Manolio TA, Burke GL, Wolfson SK Jr. Carotid-artery intima and media thickness as a risk factor for myocardial infarction and stroke in older adults. Cardiovascular Health Study Collaborative Research Group. N Engl J Med. 1999 Jan 7;340(1):14-22. doi: 10.1056/NEJM199901073400103. PMID 9878640
- [Result] Spence JD, Eliasziw M, DiCicco M, Hackam DG, Galil R, Lohmann T. Carotid plaque area: a tool for targeting and evaluating vascular preventive therapy. Stroke. 2002 Dec;33(12):2916-22. doi: 10.1161/01.str.0000042207.16156.b9. PMID 12468791
- [Result] Lorenz MW, Polak JF, Kavousi M, Mathiesen EB, Volzke H, Tuomainen TP, Sander D, Plichart M, Catapano AL, Robertson CM, Kiechl S, Rundek T, Desvarieux M, Lind L, Schmid C, DasMahapatra P, Gao L, Ziegelbauer K, Bots ML, Thompson SG; PROG-IMT Study Group. Carotid intima-media thickness progression to predict cardiovascular events in the general population (the PROG-IMT collaborative project): a meta-analysis of individual participant data. Lancet. 2012 Jun 2;379(9831):2053-62. doi: 10.1016/S0140-6736(12)60441-3. Epub 2012 Apr 27. PMID 22541275
- [Result] Polak JF, Pencina MJ, Pencina KM, O'Donnell CJ, Wolf PA, D'Agostino RB Sr. Carotid-wall intima-media thickness and cardiovascular events. N Engl J Med. 2011 Jul 21;365(3):213-21. doi: 10.1056/NEJMoa1012592. PMID 21774709
- [Result] Saba L, Saam T, Jager HR, Yuan C, Hatsukami TS, Saloner D, Wasserman BA, Bonati LH, Wintermark M. Imaging biomarkers of vulnerable carotid plaques for stroke risk prediction and their potential clinical implications. Lancet Neurol. 2019 Jun;18(6):559-572. doi: 10.1016/S1474-4422(19)30035-3. Epub 2019 Apr 4. PMID 30954372
- [Result] Lechareas S, Yanni AE, Golemati S, Chatziioannou A, Perrea D. Ultrasound and Biochemical Diagnostic Tools for the Characterization of Vulnerable Carotid Atherosclerotic Plaque. Ultrasound Med Biol. 2016 Jan;42(1):31-43. doi: 10.1016/j.ultrasmedbio.2015.09.003. Epub 2015 Oct 20. PMID 26493239
- [Result] Sakaguchi M, Kitagawa K, Nagai Y, Yamagami H, Kondo K, Matsushita K, Oku N, Hougaku H, Ohtsuki T, Masuyama T, Matsumoto M, Hori M. Equivalence of plaque score and intima-media thickness of carotid ultrasonography for predicting severe coronary artery lesion. Ultrasound Med Biol. 2003 Mar;29(3):367-71. doi: 10.1016/s0301-5629(02)00743-3. PMID 12706187